CLINICAL TRIAL: NCT05230693
Title: The SPARC App: A Smartphone Application for the Management of Sarcoidosis-Associated Fatigue
Brief Title: SPARC Smartphone Application for the Management of Sarcoidosis-Associated Fatigue
Acronym: SPARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, W. Ennis James, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00107105; 1R21EB025525 (NIH)
Record Dates: First submitted 2022-01-25; First posted 2022-02-09 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Sarcoidosis; Fatigue
MeSH Terms: conditions — Sarcoidosis; Fatigue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPARC Group (Experimental)
  Interventions: Behavioral: Sarcoidosis Patient Assessment and Resource Companion App
- Enhanced Standard Care Control Group (Active Comparator)
  Interventions: Behavioral: Enhanced Standard Care

INTERVENTIONS:
Behavioral: Sarcoidosis Patient Assessment and Resource Companion App — The first group, called the "SPARC group" will be asked to download the SPARC app onto the participant's smartphone, will be shown how to use the app, and then will be asked to use the app to do guided meditations for ten minutes twice a day
  Arms: SPARC Group
Behavioral: Enhanced Standard Care — Participants will receive education about reducing fatigue associated with sarcoidosis during a normal clinic visit.
  Arms: Enhanced Standard Care Control Group

SUMMARY:
Fatigue is a pervasive and disabling symptom in sarcoidosis with limited treatment options. There is a significant association between heightened stress and sarcoidosis-associated fatigue. The proposed project will evaluate the usability/feasibility of a smartphone-based stress management application for the self-management of sarcoidosis-associated stress and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Sarcoidosis diagnosis based on established criteria
* ≥18 years old
* able to speak, hear, and understand English
* elevated SAF (FAS score ≥22)
* owns smartphone with current data plan
* willingness and ability to use app to engage in Breathing Awareness Meditation (BAM)

Exclusion Criteria:

* history of psychotic disorder, bipolar disorder, eating disorder, narcolepsy, cancer diagnosis or treatment in past 12 months
* positive screening for potential major depression (Patient Health Questionnaire depression scale [PHQ-8; α = .86] score ≥10)
* untreated sleep apnea (based on home sleep study testing)
* sarcoidosis exacerbation in past 3 months requiring increase in sarcoidosis medications
* >2 hr travel distance to medical center (to reduce likelihood of no-show for focus groups)
* active substance abuse or binge drinking (>21 drinks/week )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SPARC Group | Enhanced Standard Care Control Group
Started | 25 | 25
Completed | 21 | 18
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Population: includes all patients who completed at least 1 month of the study
Groups:
- Total: Total of all reporting groups
Arm/Group | SPARC Group | Enhanced Standard Care Control Group | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (14.2) | 56.0 (10.7) | 54.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 6 | 10 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 8 | 14 | 22
  White | 16 | 10 | 26
  Hispanic | 1 | 0 | 1
Perceived Stress Scale (PSS-10) [Mean (Standard Deviation); unit: units on a scale] — 0-40, lower score = lower stress
  units on a scale | 19.9 (7.0) | 17.7 (6.9) | 18.5 (6.6)
Fatigue Assessment Scale [Mean (Standard Deviation); unit: units on a scale] — 0-50; higher scores = worse fatigue
  units on a scale | 30.8 (6.3) | 30.8 (7.1) | 30.8 (6.6)
King's Sarcoidosis Questionnaire [Mean (Standard Deviation); unit: units on a scale] — QOL measure, range 0(poor)-100(better)
  units on a scale | 46.5 (9.4) | 47.8 (10.7) | 47.6 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Recruited
Description: Recruitment compared to number approached
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SPARC Group | Enhanced Standard Care Control Group
Number analyzed (Participants) | 25 | 25
Participants | 25 | 25

2. Primary Outcome: Number of Participants Who Complete the Study
Description: Participants complete the study in it's entirety and are able to use the app appropriately
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- SPARC App: Intervention group
- Enhanced Standard of Care: Control group
Arm/Group | SPARC App | Enhanced Standard of Care
Number analyzed (Participants) | 25 | 24
Participants | 25 | 24

3. Primary Outcome: Number of Participants Who Maintain Adherence to at Least Daily Daily Breathing Awareness Meditation Sessions
Description: Adherence is defined by participants completing 70% of the breathing awareness meditation sessions
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Adherent: Patients in the SPARC App group that had 70% or better adherence to at least daily breathing awareness meditation
- Nonadherent: Patients in the SPARC App group that were not adherent
Arm/Group | Adherent | Nonadherent
Number analyzed (Participants) | 25 | 25
Participants | 10 | 15

4. Primary Outcome: Treatment Satisfaction
Description: System Usability Scale (SUS) consists of ten statements each with five possible answers ranging from complete rejection to complete agreement. For each statement, the participant gives his or her approval or rejection in the form of a scale ranging from 1=strong approval to 5=strong rejection. The results of the SUS questionnaire are used to calculate a numerical value (SUS score). The results can have a value between 0 (worst application imaginable) and 100 (best application imaginable)
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adherent | Nonadherent
Number analyzed (Participants) | 10 | 15
units on a scale | 60.4 (16.4) | 49.1 (15.1)

5. Secondary Outcome: Change in Sarcoidosis Associated Fatigue From Baseline to Month 6
Description: SAF is measured by Fatigue Assessment Scale which is a Fatigue Questionnaire (1 to 5-point scale x 10 questions for a total score range of 0 to 50) where a low value indicates less fatigued (better outcome) and a high value indicates more fatigued (worse outcome)
Time Frame: Week 0 and Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPARC Group | Enhanced Standard Care Control Group
Number analyzed (Participants) | 21 | 25
units on a scale | -7.1 (5.3) | 0.4 (3.8)

6. Secondary Outcome: Changes in Self-Efficacy From Baseline to Month 3
Description: Self-Efficacy is measured by the Fatigue Self-Efficacy Sale which is an 8 item scale to assess how the participant handles fatigue. Scores range from 0 to 100, with higher scores representing better fatigue self-efficacy.
Time Frame: Week 0 and Week 12
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | SPARC App | Enhanced Standard of Care
Number analyzed (Participants) | 25 | 24
score on a scale | 10.6 (20.0) | 0.6 (18.8)

7. Secondary Outcome: Changes in Stress From Baseline to Month 6
Description: Stress is measured by the Perceived Stress Scale which is a 10 item scale that asks about feelings and thoughts during the last month. The scale ranges from 0-40, lower score meaning low stress, and a higher score meaning high stress. A negative change represents an improvement (decrease) in stress
Time Frame: Week 0 and Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPARC Group | Enhanced Standard Care Control Group
Number analyzed (Participants) | 25 | 18
units on a scale | -5.0 (7.7) | -1.2 (6.3)

8. Secondary Outcome: Changes in Autonomous Motivation
Description: Autonomous motivation is measured by the Treatment Self-Regulation Questionnaire (TSRQ), which is a 15 item scale that assesses the degree of autonomous self-regulation to explain why participants engage or would engage in healthy behavior. The higher the score, the better the outcome.
Time Frame: Week 0 and Week 24
Reporting Status: Not Posted

9. Secondary Outcome: Changes in Quality of Life
Description: Quality of life is measured by the King's Sarcoidosis Health Questionnaire (KSQ), which is a 29 item scale that asks the participant questions about their general health, lung health, medications, skin, and eyes. Reliability = .90 -.97. A positive change represents an improvement (increase) in QOL. range 0-100; positive number = improvement
Time Frame: Week 0 and Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPARC Group | Enhanced Standard Care Control Group
Number analyzed (Participants) | 21 | 18
units on a scale | 11.7 (10.3) | 1.3 (9.6)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Patients were queried at month 0,1,3,6 regrading any perceived potential negative impact on the patient's health of using the smartphone app
Arm/Group | SPARC Group | Enhanced Standard Care Control Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT05230693/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT05230693/ICF_000.pdf